CLINICAL TRIAL: NCT04854876
Title: An Open-Label, Pilot Study to Evaluate the Safety, Tolerability, and Efficacy of 5-ALA-Phosphate + SFC as an Immune System Enhancer Along With Vaccination Against SARS-CoV-2 Virus Infection
Brief Title: Pilot Study to Evaluate the Safety, Tolerability, and Efficacy of 5-ALA-Phosphate + SFC as an Immune System Enhancer Along With Vaccination Against COVID-19
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The food supplement/health product registration needs to be undertaken with NHRA- Pharmaceutical Product Regulations Department
Sponsor: Royal College of Surgeons in Ireland - Medical University of Bahrain (Other)
Collaborators: Bahrain Defence Force Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BDF/R&REC/2021-566
Record Dates: First submitted 2021-04-21; First posted 2021-04-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: SARS-COV 2; Covid19
Keywords: 5-ALAPhosphate + SFC; COVID-19 Vaccination
MeSH Terms: conditions — COVID-19 | interventions — Sodium Glutamate

STUDY DESIGN:
Intervention Model Description: This is an open-label, two arm interventional exploratory study, in which one arm will consist of 100 subjects that were vaccinated with the first dose of a COVID-19 Vaccine (any brand approved in Bahrain is permitted) and those will be treated with 150mg 5-ALA Phosphate/SFC for 28 days. The second arm will consist of 100 subjects that were vaccinated with the first dose of a COVID-19 Vaccine (any brand approved in Bahrain is permitted) only (Control). This is to determine the safety and evaluate the efficacy of 5-ALA-Phosphate-SFC during the vaccination of subjects against SARS-CoV-2 (COVID-19) virus infection and to activate the immune system during SARS-CoV-2 vaccination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccinated with 1st dose of COVID-19 Vaccine & treated with 5-ALA Phosphate/SFC (Experimental): 100 subjects that were vaccinated with the first dose of a COVID-19 Vaccine (any brand approved in Bahrain is permitted) and that will be treated with 150mg 5-ALA Phosphate/SFC for 28 days
  Interventions: Dietary Supplement: 5-ALA-Phosphate + SFC (5-ALA+SFC)
- Vaccinated with 1st dose of COVID-19 Vaccine (No Intervention): 100 subjects that were vaccinated with the first dose of a COVID-19 Vaccine (any brand approved in Bahrain is permitted) only (Control)

INTERVENTIONS:
Dietary Supplement: 5-ALA-Phosphate + SFC (5-ALA+SFC) — The food supplement 5-Aminolevulinic acid phosphate and Sodium ferrous citrate (5-ALA-Phosphate + SFC) will be administered orally daily for 28 days. The dose will be in total 3 capsules of 50 mg 5-ALA-Phosphate and 28.68 mg SFC (3.04 mg as Fe) per day, 2 capsules in the morning and 1 capsule in the evening resulting in 150 mg 5-ALA-Phosphate and 86.04 mg SFC ( 9.12 mg as Fe).
  Arms: Vaccinated with 1st dose of COVID-19 Vaccine & treated with 5-ALA Phosphate/SFC

SUMMARY:
This is an open-label, two arm interventional exploratory study to evaluate the safety and efficacy of 5-ALA-Phosphate-SFC during the vaccination of subjects against SARS-CoV-2 (COVID-19) virus infection to define the safety and to activate the immune system during SARS-CoV-2 vaccination.

The primary objective of this study is to determine the safety of a 4 week daily oral administration of 5-ALA-Phosphate + SFC in subjects vaccinated with COVID-19 Vaccine

DETAILED DESCRIPTION:
This is an open-label, two arm interventional exploratory study to evaluate the safety and efficacy of 5-ALA-Phosphate-SFC during the vaccination of subjects against SARS-CoV-2 (COVID-19) virus infection to define the safety and to activate the immune system during SARS-CoV-2 vaccination.

Arm 1: 100 subjects that were vaccinated with the first dose of a COVID-19 Vaccine (any brand approved in Bahrain is permitted) and that will be treated with 150mg 5-ALA Phosphate/SFC for 28 days and

Arm 2: 100 subjects that were vaccinated with the first dose of a COVID-19 Vaccine (any brand approved in Bahrain is permitted) only (Control)

The duration of this clinical study will depend on the type of the vaccine, the subject was administered with.

Primary Endpoints: All treatment emergent AEs and SAEs Grade III and IV (CTC) with reasonable possibility of causal relationship to 5-ALA-Phosphate + SFC

Secondary Endpoint:

* Serum levels of biomarkers (CD4+/- and CD8+/- ) before and after vaccination with and without ALA/SFC administration.
* Total antibody level and neutralizing antibody level

Exploratory Endpoints:

1. Measurement of total IgA, IgM and IgG antibodies against SARS-CoV 2.
2. Measurement of neutralizing antibodies against SARS-CoV-2.

Safety:

The following safety endpoints will be assessed:

* Clinical laboratory assessments (hepatic function,)
* All reports of AEs and SAEs Grade III and IV (CTC) with reasonable possibility of causal relationship to 5-ALA-Phosphate + SFC

Efficacy:

Efficacy will be assessing the immune system related T-helper cells and antibodies after SARS-CoV-2 vaccination for each subject.

From day 0 onwards, all subjects keep a subject diary, which they fill out daily in order to record the dosage with the study treatment. Patients must meet the testing requirements on the day of the first vaccination (Day 0) and on the Day of the second vaccination and on Day 28 and on Follow-up visit.

The food supplement 5-Aminolevulinic acid phosphate and Sodium ferrous citrate (5-ALA-Phosphate + SFC) will be administered orally daily for 4 weeks at the following TOTAL daily doses:

Subjects in the vaccination + ALA/SFC arm (Arm 1) will receive:

• In total 3 capsules of 50 mg 5-ALA-Phosphate and 28.68 mg SFC (3.04 mg as Fe) per day, 2 capsules in the morning and 1 capsule in the evening resulting in 150 mg 5-ALA-Phosphate and 86.04 mg SFC ( 9.12 mg as Fe) total daily dose for 28 days

Heme is critical for appropriate oxygen binding and delivery to remote site and without the heme contained within the hemoglobin tetramer, multicellular organisms would be unable to survive. Furthermore HO-1 degrades heme into biliverdin, carbon monoxide (CO), and iron, and biliverdin is immediately reduced and turned into bilirubin by biliverdin reductase. Biliverdin/bilirubin and CO both have anti-oxidative functions and they regulate important biological processes like inflammation, apoptosis, cell proliferation, fibrosis, and angiogenesis. Therefore, HO-1 is deemed to be a promising drug target (Ryter 2006). HO-1 is a major anti-inflammatory enzyme and a key regulator that induces immune tolerance.

5-ALA-Phosphate + SFC increases heme metabolism and HO-1 via enhancement of porphyrin biology and utilizes the HO-1 for endothelial pacification strategy. Nishio reported 2014 that 5-aminolevulinic acid, a precursor of heme, in combination with divalent iron (SFC) is also able to induce HO-1 in vitro (Nishio 2014). This was attributed to the upregulation of heme synthesis and that 5-ALA+SFC transiently increased the intracellular heme amount through the phosphorylation of ERK / p38 and the nuclear translocation of a transcription factor Nrf2, as well as the depletion of a repressor protein BACH1 binding to the promoter site of HO-1. Similarly, Nakaso et al., 2003, Nishio et al., 2014, Ogawa et al., 2001, Saito et al., 2017 found that hemin administration promoted Nrf2 nuclear translocation and BACH1 dissociation leading to HO-1 induction.

Ito found in 2018 that the combination of 5-ALA 600 mg and sodium ferrous citrate (SFC) 942 mg upregulated HO-1 in PBMC at 8 h after administration while sole administration of 5-ALA or SFC was unable to induce HO-1. HO-1 in blood myeloid and plasmacytoid dendritic cells was also upregulated by the combination of 5-ALA + SFC.

In summary the versatility of the administration of 5-ALA plus iron citrate (SFC) enables the body to counteract the inflammatory reactions that the virus induces in the endothelial system and multiple organs in the event of a virus attack by increasing the formation of HO-1.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent, or with a legal representative who can provide informed consent
* Aged ≥ 21 years (at all sites)
* Subjects that have been vaccinated with the first dose of a vaccine (any brand approved in Bahrain is permitted) to protect against COVID-19 infection

Exclusion Criteria:

* Subject has acute or chronic type(s) of porphyria or a family history of porphyria.
* Subject has demonstrated previous intolerance of 5-ALA and/or SFC by topical or oral administration (except for photosensitivity)
* Pregnant or nursing women
* Males and females of reproductive potential who have not agreed to use an adequate method of contraception during the study.
* Subjects who are unable or unwilling to comply with requirements of the clinical trial.
* Participation in any other clinical trial of an experimental treatment for COVID-19
* Subjects who may be excluded at the Investigator's discretion

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
To determine the safety of a 4 week daily oral administration of 5-ALA + SFC in subject vaccinated with COVID-19 Vaccine | 28 days
  To capture the incidence of all treatment emergent AEs and SAEs Grade III and IV (CTC) with reasonable possibility of causal relationship to 5-ALA + SFC

SECONDARY OUTCOMES:
To evaluate the efficacy of 5-ALA + SFC in activating the immune system in subject vaccinated with COVID-19 Vaccine | 28 days
  To determine the serum levels of biomarkers (CD4+/- and CD8+/- ) before and after vaccination with and without 5-ALA + SFC administration and total antibody level and neutralizing antibody level

OTHER OUTCOMES:
Measurement of total IgA, IgM and IgG antibodies against SARS-CoV 2 | 28 days
  To determine measurement of total IgA, IgM and IgG antibodies against SARS-CoV 2 before and after vaccination with and without 5-ALA + SFC administration
Clinical laboratory assessments (hepatic function) | 28 days
  Monitoring of the liver enzymes before and during the study

CONTACTS AND LOCATIONS:
Overall Officials: Abdulla Darwish, Dr, Principal Investigator — Bahrain Defense Force Royal Medical Services, Military Hospital

REFERENCES:
- [Background] Ahmed R, Gray D. Immunological memory and protective immunity: understanding their relation. Science. 1996 Apr 5;272(5258):54-60. doi: 10.1126/science.272.5258.54. PMID 8600537
- [Background] Brooks A., Study 8259980 "5-ALA/SFC: A Phase I, Double-Blind, Placebo-Controlled, Single and Multiple Oral Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Caucasian and Japanese Subjects," Covance: Leeds and London, UK (2013)
- [Background] Cao WC, Liu W, Zhang PH, Zhang F, Richardus JH. Disappearance of antibodies to SARS-associated coronavirus after recovery. N Engl J Med. 2007 Sep 13;357(11):1162-3. doi: 10.1056/NEJMc070348. No abstract available. PMID 17855683
- [Background] Channappanavar R, Fett C, Zhao J, Meyerholz DK, Perlman S. Virus-specific memory CD8 T cells provide substantial protection from lethal severe acute respiratory syndrome coronavirus infection. J Virol. 2014 Oct;88(19):11034-44. doi: 10.1128/JVI.01505-14. Epub 2014 Jul 23. PMID 25056892
- [Background] Grifoni A, Weiskopf D, Ramirez SI, Mateus J, Dan JM, Moderbacher CR, Rawlings SA, Sutherland A, Premkumar L, Jadi RS, Marrama D, de Silva AM, Frazier A, Carlin AF, Greenbaum JA, Peters B, Krammer F, Smith DM, Crotty S, Sette A. Targets of T Cell Responses to SARS-CoV-2 Coronavirus in Humans with COVID-19 Disease and Unexposed Individuals. Cell. 2020 Jun 25;181(7):1489-1501.e15. doi: 10.1016/j.cell.2020.05.015. Epub 2020 May 20. PMID 32473127
- [Background] Hu X. 5-Aminolevulinic acid with sodium ferrous citrate enhance the antitumor effects of PD-L1 blockade in mouse melanoma model7th International ALA and Prophyrin Symposium (IAPS7) in Sapporo 2019.
- [Background] Ibarrondo FJ, Fulcher JA, Goodman-Meza D, Elliott J, Hofmann C, Hausner MA, Ferbas KG, Tobin NH, Aldrovandi GM, Yang OO. Rapid Decay of Anti-SARS-CoV-2 Antibodies in Persons with Mild Covid-19. N Engl J Med. 2020 Sep 10;383(11):1085-1087. doi: 10.1056/NEJMc2025179. Epub 2020 Jul 21. No abstract available. PMID 32706954
- [Background] Investigator's Brochure, SBI Pharmaceuticals Internal Document: 5-Aminolevulinic Acid (5-ALA) Phosphate Version 1.0. July, 2020
- [Background] Krammer F. SARS-CoV-2 vaccines in development. Nature. 2020 Oct;586(7830):516-527. doi: 10.1038/s41586-020-2798-3. Epub 2020 Sep 23. PMID 32967006
- [Background] Kreer C, Zehner M, Weber T, Ercanoglu MS, Gieselmann L, Rohde C, Halwe S, Korenkov M, Schommers P, Vanshylla K, Di Cristanziano V, Janicki H, Brinker R, Ashurov A, Krahling V, Kupke A, Cohen-Dvashi H, Koch M, Eckert JM, Lederer S, Pfeifer N, Wolf T, Vehreschild MJGT, Wendtner C, Diskin R, Gruell H, Becker S, Klein F. Longitudinal Isolation of Potent Near-Germline SARS-CoV-2-Neutralizing Antibodies from COVID-19 Patients. Cell. 2020 Aug 20;182(4):843-854.e12. doi: 10.1016/j.cell.2020.06.044. Epub 2020 Jul 13. PMID 32673567
- [Background] Le Bert N, Tan AT, Kunasegaran K, Tham CYL, Hafezi M, Chia A, Chng MHY, Lin M, Tan N, Linster M, Chia WN, Chen MI, Wang LF, Ooi EE, Kalimuddin S, Tambyah PA, Low JG, Tan YJ, Bertoletti A. SARS-CoV-2-specific T cell immunity in cases of COVID-19 and SARS, and uninfected controls. Nature. 2020 Aug;584(7821):457-462. doi: 10.1038/s41586-020-2550-z. Epub 2020 Jul 15. PMID 32668444
- [Background] Le TT, Cramer JP, Chen R, Mayhew S. Evolution of the COVID-19 vaccine development landscape. Nat Rev Drug Discov. 2020 Oct;19(10):667-668. doi: 10.1038/d41573-020-00151-8. No abstract available. PMID 32887942
- [Background] Long QX, Tang XJ, Shi QL, Li Q, Deng HJ, Yuan J, Hu JL, Xu W, Zhang Y, Lv FJ, Su K, Zhang F, Gong J, Wu B, Liu XM, Li JJ, Qiu JF, Chen J, Huang AL. Clinical and immunological assessment of asymptomatic SARS-CoV-2 infections. Nat Med. 2020 Aug;26(8):1200-1204. doi: 10.1038/s41591-020-0965-6. Epub 2020 Jun 18. PMID 32555424
- [Background] Matsumoto C., Study ALA-01 "Bioequivalence study of test foods A, B, and C - Based on the Plasma Concentration of 5-Aminolevulinic Acid." Kaiyu Clinic: Tokyo Japan (2010)
- [Background] Ng OW, Chia A, Tan AT, Jadi RS, Leong HN, Bertoletti A, Tan YJ. Memory T cell responses targeting the SARS coronavirus persist up to 11 years post-infection. Vaccine. 2016 Apr 12;34(17):2008-14. doi: 10.1016/j.vaccine.2016.02.063. Epub 2016 Mar 5. PMID 26954467
- [Background] Nishio Y, Fujino M, Zhao M, Ishii T, Ishizuka M, Ito H, Takahashi K, Abe F, Nakajima M, Tanaka T, Taketani S, Nagahara Y, Li XK. 5-Aminolevulinic acid combined with ferrous iron enhances the expression of heme oxygenase-1. Int Immunopharmacol. 2014 Apr;19(2):300-7. doi: 10.1016/j.intimp.2014.02.003. Epub 2014 Feb 13. PMID 24530569
- [Background] Ogawa K, Sun J, Taketani S, Nakajima O, Nishitani C, Sassa S, Hayashi N, Yamamoto M, Shibahara S, Fujita H, Igarashi K. Heme mediates derepression of Maf recognition element through direct binding to transcription repressor Bach1. EMBO J. 2001 Jun 1;20(11):2835-43. doi: 10.1093/emboj/20.11.2835. PMID 11387216
- [Background] Reed SG, Orr MT, Fox CB. Key roles of adjuvants in modern vaccines. Nat Med. 2013 Dec;19(12):1597-608. doi: 10.1038/nm.3409. Epub 2013 Dec 5. PMID 24309663
- [Background] Ripperger T. J. et al., Detection, prevalence, and duration of humoral responses to SARS-CoV-2 under conditions of limited population exposure. medRxiv, (2020).
- [Background] Rodda LB, Netland J, Shehata L, Pruner KB, Morawski PA, Thouvenel CD, Takehara KK, Eggenberger J, Hemann EA, Waterman HR, Fahning ML, Chen Y, Hale M, Rathe J, Stokes C, Wrenn S, Fiala B, Carter L, Hamerman JA, King NP, Gale M Jr, Campbell DJ, Rawlings DJ, Pepper M. Functional SARS-CoV-2-Specific Immune Memory Persists after Mild COVID-19. Cell. 2021 Jan 7;184(1):169-183.e17. doi: 10.1016/j.cell.2020.11.029. Epub 2020 Nov 23. PMID 33296701
- [Background] Ryter SW, Alam J, Choi AM. Heme oxygenase-1/carbon monoxide: from basic science to therapeutic applications. Physiol Rev. 2006 Apr;86(2):583-650. doi: 10.1152/physrev.00011.2005. PMID 16601269
- [Background] Saito K, Fujiwara T, Ota U, Hatta S, Ichikawa S, Kobayashi M, Okitsu Y, Fukuhara N, Onishi Y, Ishizuka M, Tanaka T, Harigae H. Dynamics of absorption, metabolism, and excretion of 5-aminolevulinic acid in human intestinal Caco-2 cells. Biochem Biophys Rep. 2017 Jul 13;11:105-111. doi: 10.1016/j.bbrep.2017.07.006. eCollection 2017 Sep. PMID 28955775
- [Background] Schmidt ME, Varga SM. The CD8 T Cell Response to Respiratory Virus Infections. Front Immunol. 2018 Apr 9;9:678. doi: 10.3389/fimmu.2018.00678. eCollection 2018. PMID 29686673
- [Background] Tang F, Quan Y, Xin ZT, Wrammert J, Ma MJ, Lv H, Wang TB, Yang H, Richardus JH, Liu W, Cao WC. Lack of peripheral memory B cell responses in recovered patients with severe acute respiratory syndrome: a six-year follow-up study. J Immunol. 2011 Jun 15;186(12):7264-8. doi: 10.4049/jimmunol.0903490. Epub 2011 May 16. PMID 21576510
- [Background] Vartak A, Sucheck SJ. Recent Advances in Subunit Vaccine Carriers. Vaccines (Basel). 2016 Apr 19;4(2):12. doi: 10.3390/vaccines4020012. PMID 27104575
- [Background] Zhao J, Zhao J, Mangalam AK, Channappanavar R, Fett C, Meyerholz DK, Agnihothram S, Baric RS, David CS, Perlman S. Airway Memory CD4(+) T Cells Mediate Protective Immunity against Emerging Respiratory Coronaviruses. Immunity. 2016 Jun 21;44(6):1379-91. doi: 10.1016/j.immuni.2016.05.006. Epub 2016 Jun 7. PMID 27287409
- [Background] Zhao J, Zhao J, Perlman S. T cell responses are required for protection from clinical disease and for virus clearance in severe acute respiratory syndrome coronavirus-infected mice. J Virol. 2010 Sep;84(18):9318-25. doi: 10.1128/JVI.01049-10. Epub 2010 Jul 7. PMID 20610717
- [Background] Bilich T., Nelde A., Heitmann J.S., Maringer Y., Roerden M., Bauer J., Rieth J., Wacker M., Peter A., Hörber S., Rachfalski D., Märklin M., Stevanovic A., Rammensee G., Salih H.R., Walz J.S. Differential kinetics of T cell and antibody responses delineate dominant T cell epitopes in long-term immunity after COVID-19, DOI: https://doi.org/10.21203/rs.3.rs-114499/v1